CLINICAL TRIAL: NCT04301674
Title: Pilot Study of Metabolomics in Occupational Asthma
Brief Title: Metabolomics in Occupational Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Owlstone Ltd (Industry)
Responsible Party: Principal Investigator, Bato Hammarstrøm, Senior consultant/Research group leader, Oslo University Hospital
Other Study IDs: UO1
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Asthma, Occupational
MeSH Terms: conditions — Asthma, Occupational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Volatile Organic Compounds (VOC) in exhaled air
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Occupational Asthma: Patients refered for assesment of occupational asthma
  Interventions: Device: Breath Biopsy
- Respiratory Healthy Control: Employees at Oslo University Hospital
  Interventions: Device: Breath Biopsy

INTERVENTIONS:
Device: Breath Biopsy — ReCIVA breath sampler (Owlstone Medical, Cambridge, UK)

SUMMARY:
The project aims to increase the diagnostic accuracy in occupational asthma (OA), with emphasis on Irritant Induced Asthma (IIA). Currently, most patients are evaluated in occupational medicine by comparing the exposure and symptom characteristics with epidemiological data. Biological markers may be present in AA, but presently not in IIA. The majority of cases evaluated are considered as possible IIA, i.e. low-dose multiple exposures. VOC features will be analyzed with the Breath Biopsy® and TD-GS-MS (Owlstone Medical Ltd, UK).

ELIGIBILITY:
Inclusion Criteria:

* capable of informed consent.
* asthma diagnosis established by lung specialist or healthy control.

Exclusion Criteria:

* skin allergy towards plastics or rubber.
* immunocompromised by oral medication.
* contagious respiratory disease.
* biopsy of lung parenchyma within the last 36 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with occupational asthma, referred to the Unit of Environmental and Occupational medicine OUS for evaluation of OA.and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Discovery of VOC Biomarkers in Asthma | Baseline
  To evaluate the sensitivity, specificity, positive and negative predictive value of VOC biomarkers in exhaled breath samples to identify asthma.
Discovery of VOC Biomarkers in Occupational Irritant Asthma | Baseline
  To evaluate the sensitivity, specificity, positive and negative predictive value of VOC biomarkers in exhaled breath samples to identify irritant asthma after occupational exposures.

CONTACTS AND LOCATIONS:
Overall Officials: Bato Hammarstrøm, MD/PhD, Principal Investigator — Oslo University Hospital; Tonje Trulssen Hildre, M.Sc., Study Chair — Oslo University Hospital; Hilde Heiro, MD, Study Chair — Oslo University Hospital; Britt G Randem, MD/PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No